CLINICAL TRIAL: NCT04406168
Title: Assessment of Urinary Diversions Outcomes Post Radical Cystectomy in Asyut University Urology Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Mahmoud Abdellah, resident of urology, Assiut University
Other Study IDs: urinary diversions outcomes
Record Dates: First submitted 2020-05-10; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Urinary Diversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: urinary diversion — follow up outcomes of urinary diversion

SUMMARY:
Radical cystectomy (RC) for bladder cancer requires reconstruction of the lower urinary tract. Both continent and incontinent diversions are available for urinary reconstruction after RC. Types of urinary diversions include ( ileal conduit, uretero-cutaneous, ureterosigmoidostomy and orthotopic bladder) The decision process is complex and involves consideration of issues related to cancer stage, patient comorbidities, treatment needs, and patient desires related to Quality of life and intraoperative findings. Outcomes of urinary diversions include 1- survival rate (cancer specific or overall survival). 2- Oncological failure (local, distant or LNs). 3- Complications (perioperative, intraoperative or post-operative).

In this study, all these outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* * All patients underwent radical cystectomy more than 1 year

Exclusion Criteria:

* incomplete data
* patients underwent RC outside urology department and presented for treatment of complications.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All cases that fulfil the selection criteria that have been admitted in Asyut university urology hospital (non probability sample size) with expected size of 40 patients starting from 01/01/2013 to1/05/2020.
  Additionally, the competence of follow-up will be approved by imaging and medical records.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients presented by complications | 1 year post operative
  such as (change from baseline of the SCR - urinary tract infections - stone formation - stricture at site of anastomosis or stromal stenosis )
Rate of patients developed recurrence | 1 year post operative
  recurrence of cancer
Survival rate (overall survival & cancer specific) | 1 year post operative
  patient live post operative

CONTACTS AND LOCATIONS:
Overall Officials: salah s abdelhafez, Study Director — prof
Locations (1):
- Assiut University, Asyut, Elgam3a, Egypt

IPD SHARING:
Plan to Share IPD: Undecided